CLINICAL TRIAL: NCT07183605
Title: Central Catheter Anti-Xa Sampling Study for Accurate aNalysis and Reliable Dosage Assessment
Brief Title: Comparison of Heparin Anti-Xa Activity From Central Venous Catheter Samples Using a 5 mL Syringe Flush or a Vacuum Tube Flush Versus Peripheral Vein Samples in ICU Patients
Acronym: CASSANDRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUO-2024-27
Record Dates: First submitted 2025-08-29; First posted 2025-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anticoagulants and Bleeding Disorders
Keywords: Unfractionated Heparin; Anti-Xa Activity; Catheterization, Central Venous; Blood Specimen Collection; Intensive care
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence A, B, A, B (Experimental): First and third samples with syringe flush; second and fourth with vacuum tube flush
  Interventions: Procedure: catheter flushing techniques
- Sequence A, B, B, A (Experimental): First and fourth samples with syringe flush; second and third with vacuum tube flush
  Interventions: Procedure: catheter flushing techniques
- Sequence B, A, B, A (Experimental): Second and fourth samples with syringe flush; first and third with vacuum tube flush
  Interventions: Procedure: catheter flushing techniques
- Sequence B, A, A, B (Experimental): Second and third samples with syringe flush; first and fourth with vacuum tube flush
  Interventions: Procedure: catheter flushing techniques

INTERVENTIONS:
Procedure: catheter flushing techniques — Two catheter flushing techniques will be compared:
  * Method A: A 5 mL flush performed with a syringe over 5 seconds.
  * Method B: A 5 mL flush using a vacuum tube (standard discard tube).

SUMMARY:
The goal is to investigate whether blood samples drawn from a central venous catheter can provide reliable measurements of unfractionated heparin (UFH) anti-Xa activity, compared to the standard method of peripheral vein puncture, in intensive care unit (ICU) patients receiving continuous intravenous UFH.

To evaluate the reliability of central venous blood sampling, the study will compare anti-Xa activity levels obtained simultaneously from two different types of blood draws: one from a peripheral vein (reference method), and the other from the central line using one of two flushing techniques.

The two central flushing techniques being studied are:

* A 5 mL syringe flush performed over 5 seconds, followed by blood collection.
* A vacuum tube flush that draws and discards 5 mL of blood, followed by blood collection.

Each patient will undergo four pairs of simultaneous blood draws, using both central techniques in a randomized sequence. The main objective is to assess whether the anti-Xa levels from central samples are equivalent to those from peripheral vein puncture, with a predefined margin of equivalence of ±0.05 IU/mL.

Findings from this study may support the use of central venous catheters for routine anti-Xa monitoring in ICU patients, potentially avoiding painful or technically difficult peripheral vein punctures.

DETAILED DESCRIPTION:
Unfractionated heparin (UFH) is widely used in intensive care units (ICUs) and requires close monitoring, most commonly through the measurement of anti-Xa activity.

The reference method for anti-Xa monitoring involves blood sampling by peripheral vascular puncture. However, in ICU patients, peripheral access may be challenging or painful, and central venous catheters are often available and already used for UFH infusion. Sampling from these central lines could be a convenient alternative, but residual heparin in the catheter may contaminate the sample, leading to falsely elevated anti-Xa results.

The CASSANDRA study (Central catheter Anti-Xa Sampling Study for Accurate aNalysis and Reliable Dosage Assessment) is a prospective, monocentric, comparative study designed to assess whether anti-Xa activity levels obtained from central venous catheter samples are equivalent to those from peripheral vein samples.

To be eligible for inclusion, patients must already have a central venous catheter in place and require continuous intravenous unfractionated heparin administration through the distal lumen of the central venous catheter.

A three-way stopcock will be placed upstream of the infusion tubing to allow temporary interruption of UFH infusion during sampling.

Two catheter flushing techniques will be compared:

* Method A: A 5 mL flush performed with a syringe over 5 seconds.
* Method B: A 5 mL flush using a vacuum tube (standard discard tube).

For each patient, four pairs of simultaneous blood samples will be collected, according to a randomized sequence alternating between methods A and B. In each pair, one sample will be drawn from the central venous catheter and the other from a fresh peripheral vein puncture (reference). All anti-Xa assays will be performed, but only the results from peripheral vein samples (reference method) will be made available to clinicians. Anti-Xa results from central venous catheter samples will remain blinded to the clinical team to avoid influencing patient management.

The primary outcome is the absolute difference in anti-Xa activity between central venous catheter samples (either method) and peripheral samples. Equivalence is defined as a mean difference not exceeding 0.05 IU/mL. Secondary outcomes include Bland-Altman agreement limits between each central method and the peripheral reference.

Results of this study may support the safe use of central venous sampling for routine anti-Xa monitoring in ICU patients, provided an appropriate flushing method is used.

ELIGIBILITY:
Inclusion Criteria:

* Person (or support person/relative if unable to do so) who has agreed to participate in the study
* 18 years of age or older
* Hospitalized in intensive care medicine
* Having a central venous catheter with at least three lumens (internal jugular, subclavian or femoral) already in place
* Receiving continuous intravenous unfractionned heparin, with target Anti-Xa activity between 0.3 and 0.7 IU/ml.

Exclusion Criteria:

* Protected person (under guardianship or curatorship)
* Person under court protection
* Person deprived of liberty
* Person not affiliated to the French social security
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Difference in anti-Xa activity values between the two sampling sites. | From inclusion to the four pairs of simultaneous blood samples collected assessed up to Day 28
  Difference in anti-Xa activity values between the two sampling sites: central venous catheter with a 5 mL discard using either a syringe or a vacuum tube, versus peripheral vein puncture, the latter being considered the reference method.
  Equivalence is defined a priori as a mean absolute difference not exceeding 0.05 IU/mL of anti-Xa activity.

SECONDARY OUTCOMES:
Equivalence of anti-Xa activity measurements between central venous catheter sampling using flush method A (5 mL syringe discard) and peripheral vein puncture. | From inclusion to the four pairs of simultaneous blood samples collected assessed up to Day 28
  Agreement limits of anti-Xa activity measurements between central venous catheter sampling using flush method A and peripheral vein puncture.
Equivalence of anti-Xa activity measurements between central venous catheter sampling using flush method B (5 mL vacuum tube discard) and peripheral vein puncture. | From inclusion to the four pairs of simultaneous blood samples collected assessed up to Day 28
  Agreement limits of anti-Xa activity measurements between central venous catheter sampling using flush method B and peripheral vein puncture.
  In both cases, the anti-Xa activity measured from the peripheral vein is considered the reference

OTHER OUTCOMES:
Types and durations of organ support therapies | From enrollment to Day 28 or discharge (whichever comes first)
  Organ support requirements, including number of days on mechanical ventilation, renal replacement therapy, or extracorporeal membrane oxygenation (ECMO).
Thromboembolic and bleeding complications | From enrollment to Day 28 or discharge (whichever comes first)
  Description of thrombotic and bleeding complications during the ICU stay, with bleeding events graded according to ISTH severity criteria.
Types of blood products transfused | From enrollment to Day 28 or discharge (whichever comes first)
  Type of blood products transfused (red blood cells, frozen plasma, platelets) during the ICU stay will be recorded.
Number of blood products transfused | Day 28 or discharge (whichever comes first)
  Number of blood products transfused during the ICU stay.
Volumes of blood products transfused | Day 28 or discharge (whichever comes first)
  Volume of blood products transfused during the ICU stay.
Inflammatory status, as reflected by fibrinogen levels. | Day 28 or discharge (whichever comes first)
  Fibrinogen level
Inflammatory status, as reflected by platelet levels. | Day 28 or discharge (whichever comes first)
  Platelets count
Total dose of protamine administered during the ICU stay | Day 28 or discharge (whichever comes first)
Hemoglobin variations during the ICU stay | Day 28 or discharge (whichever comes first)
Number and values of anti-Xa UFH assays performed | Day 28 or discharge (whichever comes first)
Vital status at ICU discharge | Up to 6 months
  Vital status (alive or deceased) assessed at the time of intensive care unit (ICU) discharge, based on the final medical record and discharge summary.
Number of discrepancies between therapeutic actions | From inclusion to Day 28
  Comparison of the number of discrepancies between therapeutic actions (i.e., heparin dose adjustments based on the unit's therapeutic protocol) undertaken in response to anti-Xa results obtained from the reference method (peripheral vein puncture) and those that would have been undertaken if anti-Xa results from central venous catheter samples had been used.
Reason for ICU admission | From enrollment to Day 28 or discharge (whichever comes first)
  Descriptive classification of the primary reason for ICU admission, based on the initial diagnosis recorded in the patient's medical chart at inclusion.
Indication for anticoagulation | From enrollment to Day 28 or discharge (whichever comes first)
  Descriptive classification of the medical indication for initiating therapeutic anticoagulation with unfractionated heparin (e.g., venous thromboembolism, atrial fibrillation, extracorporeal support, etc.) as recorded at ICU admission.
Types and durations of organ support therapies | From enrollment to Day 28 or discharge (whichever comes first)
  Number of days each organ support therapy was used during the ICU stay, including mechanical ventilation, renal replacement therapy, vasopressors, or extracorporeal membrane oxygenation (ECMO), as documented in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire MULLER, Dr, Principal Investigator — CHU Orléans
Locations (1):
- Chu Orleans, Orléans, France